CLINICAL TRIAL: NCT06144216
Title: Scaling Up Trauma-Informed Outreach with People Affected by Violence
Brief Title: Scaling Up Trauma-Informed Outreach with People Affected by Violence - CLOE Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other); Michael Smith Health Research BC (Unknown); University of Windsor (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Victoria Bungay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H23-02810; H24-01477
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gender-based Violence; Outreach Intervention
Keywords: Gender-based Violence; Outreach Intervention; Trauma-informed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLOE Outreach Intervention (Experimental): Participants enrolled in CLOE intervention
  Interventions: Other: CLOE Outreach Intervention

INTERVENTIONS:
Other: CLOE Outreach Intervention — The CLOE outreach intervention is a community-led, strengths-based, and trauma-informed program to support self-identifying women and youth who experience interpersonal and structural gender-based violence. Outreach services are designed to mitigate the effects of gender-based violence, build trusting relationships with service providers, and improve safety, well-being and engagement with health and social care.

SUMMARY:
This mixed methods, community-based study examines the implementation and outcomes of the Community-Led Outreach and Engagement Model (CLOE) for women and youth affected by violence. Outreach services are designed to mitigate the effects of gender-based violence, build trusting relationships with service providers, and improve safety, well-being and engagement with health and social care. Over a 2-year implementation period, we will test how outreach, combined with enhanced service integration, supports participants to identify priority needs and can bridge the gap in accessible and appropriate service with people affected by violence.

DETAILED DESCRIPTION:
Using community-based participatory research approaches, we implement and test an empirically driven model of outreach with people affected by violence to determine the effectiveness of the model for participants' trust in service providers, safety, and access to appropriate health and social care. The study represents a community-academic partnership between the PI, co-applicants and the Central Okanagan Elizabeth Fry Society (COEFS) and the Welcome Centre Shelter for Women and Families.

There are 4 primary research questions:

1. How effective is the intervention to achieve participant trust in the outreach service program?
2. How effective is the outreach intervention in facilitating participant connection to (a) health services; (b) social services; and (c) legal services?
3. How effective is the outreach intervention in achieving participant safety plans for (a) material, (b) psychological and (c) physical safety?
4. What are the environmental factors that enable or confound the success of the outreach intervention to achieve effectiveness for (a) trust, (b) service connections and (c) safety?

Research Method:

This study is part of a broader program of research utilizing a case-based, intervention study design that employs mixed methods of both quantitative and qualitative data. The outreach intervention consists of 1-1 outreach service provided by trained outreach interventionists to enrolled and consented participants.

Participants will be assigned an outreach interventionist for a one year period. During this time, interventionists and participants will complete a strengths-based assessment to identify participants' current resources and the types of health and social support (e.g., housing, legal, health care access, financial assistance) required. The interventionist and participant will then co-develop a plan to prioritize needs and work collaboratively to address these needs. Plans and progress will be documented by the interventionist in a participant file. Surveys will be conducted at baseline and 4 month intervals by a trained research assistant to measure changes over time in core outcome measures associated with this study (e.g., trust, safety planning, attainment of priority needs). 1-1 qualitative interviews will be conducted at time point 12 months to enable richer understanding of the factors influencing intervention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* have been referred to community partner organization for services
* able to communicate in English
* age 12-18 (gender inclusive)
* 19 years or older (self-identifying women)

Exclusion Criteria:

* Self-identifying men 19 years or older who experience violence will be excluded as the study aims to address gender-based violence with self-identifying women and youth (as per the funded SSHRC grant objectives). Community partner organizations will enable referral for any men to appropriate services.
* People who do not have a referral for service delivery within the two community partner organizations.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Youth (ages 12-18) of all genders, self-identifying women 19 & over
Enrollment: 400 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in trust from baseline to 4 months | Baseline & 4 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 4 months post-baseline
Change in trust from baseline to 8 months | Baseline & 8 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 8 months post-baseline
Change in trust from baseline to 12 months | Baseline & 12 months
  Change in trust achieved by the program with participants, measured using participants' self-rated trust in program rated from 1 to 5, with higher scores indicating higher trust and comparing baseline to 12 months post-baseline
Safety in home setting at baseline | Baseline
  Self-reported safety in current home setting using a rating of 1 to 5 with higher scores being higher safety
Safety in home setting at 4 months | 4 months post-baseline
  Self-reported safety in current home setting using a rating of 1 to 5 with higher scores being higher safety
Safety in home setting at 8 months | 8 months post-baseline
  Self-reported safety in current home setting using a rating of 1 to 5 with higher scores being higher safety
Safety in home setting at 12 months | 12 months post-baseline
  Self-reported safety in current home setting using a rating of 1 to 5 with higher scores being higher safety
Safety in community setting at baseline | Baseline
  Self-reported safety in community using a rating of 1 to 5 with higher scores being higher safety
Safety in community setting at 4 months | 4 months post-baseline
  Self-reported safety in community using a rating of 1 to 5 with higher scores being higher safety
Safety in community setting at 8 months | 8 months post-baseline
  Self-reported safety in community using a rating of 1 to 5 with higher scores being higher safety
Safety in community setting at 12 months | 12 months post-baseline
  Self-reported safety in community using a rating of 1 to 5 with higher scores being higher safety
Safety in health care encounters at baseline | Baseline
  Self-reported safety in clinical and health care encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in health care encounters at 4 months | 4 months post-baseline
  Self-reported safety in clinical and health care encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in health care encounters at 8 months | 8 months post-baseline
  Self-reported safety in clinical and health care encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in health care encounters at 12 months | 12 months post-baseline
  Self-reported safety in clinical and health care encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in socio-legal service encounters at baseline | Baseline
  Self-reported safety in socio-legal service encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in socio-legal service encounters at 4 months | 4 months post-baseline
  Self-reported safety in socio-legal service encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in socio-legal service encounters at 8 months | 8 months post-baseline
  Self-reported safety in socio-legal service encounters using a rating of 1 to 5 with higher scores being higher safety
Safety in socio-legal service encounters at 12 months | 12 months post-baseline
  Self-reported safety in socio-legal service encounters using a rating of 1 to 5 with higher scores being higher safety

SECONDARY OUTCOMES:
Program facilitates connection to services from baseline to 4 months | Baseline & 4 months
  Connection to services facilitated by outreach intervention, measured using participants' self-assessment of services needed and ability to connect (yes/no)
Program facilitates connection to services from baseline to 8 months | Baseline & 8 months
  Connection to services facilitated by outreach intervention, measured using participants' self-assessment of services needed and ability to connect (yes/no)
Program facilitates connection to services from baseline to 12 months | Baseline & 12 months
  Connection to services facilitated by outreach intervention, measured using participants' self-assessment of services needed and ability to connect (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bungay, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No